CLINICAL TRIAL: NCT01466660
Title: LUX-Lung 7: A Randomised, Open-label Phase IIb Trial of Afatinib Versus Gefitinib as First-line Treatment of Patients With EGFR Mutation Positive Advanced Adenocarcinoma of the Lung
Brief Title: LUX-Lung 7: A Phase IIb Trial of Afatinib(BIBW2992) Versus Gefitinib for the Treatment of 1st Line EGFR Mutation Positive Adenocarcinoma of the Lung
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200.123; 2011-001814-33 (EudraCT Number)
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — Afatinib; Gefitinib

ARMS (2):
- afatinib (Experimental): afatinib once daily.
  Interventions: Drug: Afatinib
- gefitinib (Active Comparator): gefitinib once daily
  Interventions: Drug: gefitinib

INTERVENTIONS:
Drug: Afatinib — afatinib once daily
  Other Names: Giotrif® / Gilotrif®
  Arms: afatinib
Drug: gefitinib — Gefitinib once daily
  Arms: gefitinib

SUMMARY:
This is a randomised, open-label, phase IIb trial of afatinib to compare to gefitinib in first-line treatment setting with patients who are having epidermal growth factor receptor mutation positive advanced adenocarcinoma of the lung.

ELIGIBILITY:
Inclusion criteria:

1. Pathologically confirmed diagnosis of Stage IIIB / IV adenocarcinoma of the lung.
2. Documented activating epidermal growth factor receptor mutation (Del19 and/or L858R) with tumour tissues.
3. At least one measurable lesion according to response evaluation criteria in solid tumours version 1.1
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
5. Age >= 18 years.
6. Adequate organ function as defined by the following criteria:

Serum aspartate transaminase(AST) and serum alanine transaminase(ALT) =< 3 x upper limit of normal (ULN), or AST and ALT =<5 x ULN if liver function abnormalities are due to underlying malignancy Total serum bilirubin =<1.5 x ULN Absolute neutrophil count (ANC) >=1.5 x 109/L Creatinine clearance > 45ml / min Platelets >= 75 x 109/L

Exclusion criteria:

1. Prior systemic chemotherapy for stage IIIB or IV non-small cell lung cancer. Neo-/adjuvant chemotherapy, chemoradiation or radiotherapy is permitted if at least 12 months has elapsed prior to disease progression.
2. Prior treatment with epidermal growth factor receptor targeting small molecules or antibodies.
3. Major surgery within 4 weeks of study randomisation.
4. Active brain metastases
5. Meningeal carcinomatosis.
6. Previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured in the opinion of investigator.
7. Known pre-existing interstitial lung disease.
8. Clinically relevant cardiovascular abnormalities as judged by the investigator.
9. Cardiac left ventricular function with resting ejection fraction of less than institutional lower limit of normal.
10. Women of child-bearing potential (WOCBP) and men who are able to father a child, unwilling to be abstinent or use adequate contraception prior to study entry, for the duration of study participation and for at least 2 months after treatment has ended.
11. Pregnancy or breast-feeding.
12. Active hepatitis and/or known HIV carrier
13. Any prohibited concomitant medications for therapy with afatinib or gefitinib

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2011-12-13 (Actual); Primary Completion 2016-04-08 (Actual); Study Completion 2019-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (63):
- Australia (7):
  - Chris Obrien Lifehouse, Camperdown, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Haematology & Oncology Clinics of Australasia (HOCA), South Brisbane, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Austin Health, Heidelberg, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Canada (6):
  - Cross Cancer Institute (University of Alberta), Edmonton, Alberta
  - British Columbia Cancer Agency (BCCA) - Fraser Valley Cancer, Surrey, British Columbia
  - BC Cancer Agency - Vancouver, Vancouver, British Columbia
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Montreal General Hospital - McGill University Health Centre, Montreal, Quebec
- China (7):
  - Cancer Hospital of Chinese Academy of Medical Science, Beijing
  - Beijing Cancer Hospital, Beijing
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - The Affiliated Cancer Hospital, Guangxi Medical University, Nanning
  - Shanghai Chest Hospital, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - The First Hospital of Chinese Medical University, Shenyang
- France (8):
  - CTR Oncologie du Pays Basque, Onco, Bayonne, Bayonne
  - CTR François Baclesse, Caen
  - HOP Intercommunal, Créteil
  - HOP Michallon, La Tronche
  - HOP Dupuytren 1, Limoges
  - CTR Leon Berard, Lyon
  - CTR René Gauducheau, Saint-Herblain
  - HOP Sud-Réunion, Pneumo, Saint Pierre, St-Pierre - La Réunion
- Germany (3):
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
- Ireland (2):
  - St James's Hospital, Dublin
  - Beaumont Hospital, Dublin
- Oslo Universitetssykehus HF, Radiumhospitalet, Oslo, Norway
- Singapore (2):
  - National Cancer Centre, Singapore
  - Johns Hopkins Singapore International Medical Center, Singapore
- South Korea (6):
  - Chungbuk National University Hospital, Cheongju-si
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (5):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Central de Asturias, Oviedo
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Virgen del Rocío, Seville
- Sweden (4):
  - Sahlgrenska US, Göteborg, Gothenburg
  - Universitetssjukhuset, Linköping, Linköping
  - Skånes universitetssjukhus, Lund, Lund
  - Karolinska Univ. sjukhuset, Stockholm
- Taiwan (5):
  - Taichung Veterans General Hospital, Taichung
  - NCKUH, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipe Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital(Linkou), Taoyuan District
- United Kingdom (5):
  - Aberdeen Royal Infirmary, Aberdeen
  - Birmingham City Hospital, Birmingham
  - Velindre Cancer Centre, Cardiff
  - Western General Hospital, Edinburgh
  - Royal Surrey County Hospital, Guildford

REFERENCES:
- [Derived] Wu YL, Sequist LV, Tan EH, Geater SL, Orlov S, Zhang L, Lee KH, Tsai CM, Kato T, Barrios CH, Schuler M, Hirsh V, Yamamoto N, O'Byrne K, Boyer M, Mok T, Peil B, Marten A, Chih-Hsin Yang J, Paz-Ares L, Park K. Afatinib as First-line Treatment of Older Patients With EGFR Mutation-Positive Non-Small-Cell Lung Cancer: Subgroup Analyses of the LUX-Lung 3, LUX-Lung 6, and LUX-Lung 7 Trials. Clin Lung Cancer. 2018 Jul;19(4):e465-e479. doi: 10.1016/j.cllc.2018.03.009. Epub 2018 Mar 17. PMID 29653820
- [Derived] Paz-Ares L, Tan EH, O'Byrne K, Zhang L, Hirsh V, Boyer M, Yang JC, Mok T, Lee KH, Lu S, Shi Y, Lee DH, Laskin J, Kim DW, Laurie SA, Kolbeck K, Fan J, Dodd N, Marten A, Park K. Afatinib versus gefitinib in patients with EGFR mutation-positive advanced non-small-cell lung cancer: overall survival data from the phase IIb LUX-Lung 7 trial. Ann Oncol. 2017 Feb 1;28(2):270-277. doi: 10.1093/annonc/mdw611. PMID 28426106
- [Derived] Park K, Tan EH, O'Byrne K, Zhang L, Boyer M, Mok T, Hirsh V, Yang JC, Lee KH, Lu S, Shi Y, Kim SW, Laskin J, Kim DW, Arvis CD, Kolbeck K, Laurie SA, Tsai CM, Shahidi M, Kim M, Massey D, Zazulina V, Paz-Ares L. Afatinib versus gefitinib as first-line treatment of patients with EGFR mutation-positive non-small-cell lung cancer (LUX-Lung 7): a phase 2B, open-label, randomised controlled trial. Lancet Oncol. 2016 May;17(5):577-89. doi: 10.1016/S1470-2045(16)30033-X. Epub 2016 Apr 12. PMID 27083334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two-arm, randomised (1:1 ratio), open-label, parallel group trial.
  In the study disease response was assessed by Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Afatinib: Afatinib film-coated tablets administered orally, once daily. Starting dose was 40 milligram (mg), dose escalation to 50mg was allowed after completing one 28-day treatment course, dose reduction to 40mg, 30mg or 20mg was required in the presence of protocol-defined adverse events. Continuous daily dosing until disease progression, occurrence of unacceptable adverse events, or other reason necessitating withdrawal.
- Gefitinib: Gefitinib film-coated tablets, administered orally, once daily. Starting dose was 250mg, the investigator was allowed to modify dosing in the presence of drug-related adverse events. Continuous daily dosing until disease progression, occurrence of unacceptable adverse events, or other reason necessitating withdrawal.
Period: Overall Study
Arm/Group | Afatinib | Gefitinib
Started | 160 | 159
Completed | 0 (On treatment at analysis cut-off date, 12 April 2019) | 0 (On treatment at analysis cut-off date, 12 April 2019)
Not Completed | 160 | 159
Not completed — Progressive Disease (RECIST 1.1) | 120 | 127
Not completed — Worsening of underlying cancer disease | 5 | 2
Not completed — Other adverse event | 19 | 18
Not completed — Protocol Violation | 2 | 1
Not completed — Refused continuation of trial medication | 4 | 3
Not completed — Other reason not defined above | 10 | 8

BASELINE CHARACTERISTICS:
Population: Randomised set which included all patients randomised to receive treatment, whether treated or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib | Gefitinib | Total
Number analyzed (Participants) | 160 | 159 | 319
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (11.5) | 63.0 (10.4) | 62.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 106 | 197
  Male | 69 | 53 | 122
Race (NIH/OMB) [Count of Participants; unit: Participants] — "Unknown or Not Reported" reflects the participants in France where race was not recorded.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 94 | 88 | 182
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 0 | 1
    White | 48 | 54 | 102
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 17 | 17 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) defined as the time from date of randomisation to date of disease progression, or date of death if a patient died earlier. Participants with no event (Disease progression (PD) or death) were censored. PD was primarily evaluated for the primary analysis by an independent central imaging review according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1. Per RECIST version 1.1. for target lesions and assessed by Computed Tomography (CT)-scan or Magnetic Resonance Imaging (MRI): PD, At least a 20% increase in the sum of the longest diameter (SoD) of target lesions taking as reference the smallest SoD of target lesions recorded since the treatment started, together with an absolute increase in the SoD of target lesions of at least 5 millimetre (mm) or the appearance of one or more new lesions. For the final analysis (analysis cut-off date 12 April 2019) status and date of PD were determined by investigator assessment.
Time Frame: From first drug administration until 28 days after last drug administration + Follow-Up period for collecting information on disease progression or death, up to 2465 days.
Population: Randomised set which included all patients randomised to receive treatment, whether treated or not.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib | Gefitinib
Number analyzed (Participants) | 160 | 159
Months | 12.78 [10.91 to 14.72] | 11.17 [9.49 to 12.81]
Statistical Analysis 1: Comparison: Afatinib vs Gefitinib; Exploratory trial, no formal hypotheses were tested; Test type: Superiority or Other; p = 0.0891, Log Rank — p-value was not adjusted for multiple comparisons; Stratified by Epidermal Growth Factor Receptor (EGFR) mutation group and presence of brain metastases at baseline; Hazard Ratio (HR) = 0.822, 95% CI 2-sided [0.655 to 1.032] — A Cox proportional hazards model, stratified by EGFR mutation group and presence of baseline brain metastases was used to estimate the hazard ratio calculated as Afatinib divided by Gefitinib

2. Primary Outcome: Time to Treatment Failure (TTF) (Main Overall Survival Analysis Cut-off Date, 08 April 2016)
Description: Time to Treatment Failure (TTF) which was the time from the date of randomisation to the date of i.e. permanent treatment discontinuation for any reason.
Time Frame: From first drug administration until last drug administration, up to 1482 days
Population: Randomised set which included all patients randomised to receive treatment, whether treated or not.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib | Gefitinib
Number analyzed (Participants) | 160 | 159
Months | 13.67 [11.89 to 14.95] | 11.53 [10.09 to 13.11]
Statistical Analysis 1: Comparison: Afatinib vs Gefitinib; Exploratory trial, no formal hypotheses were tested; Test type: Superiority or Other; p = 0.0136, Log Rank — p-value was not adjusted for multiple comparisons; Stratified by EGFR mutation group and presence of brain metastases at baseline; Hazard Ratio (HR) = 0.750, 95% CI 2-sided [0.595 to 0.944] — Ratio calculated as Afatinib divided by Gefitinib

3. Primary Outcome: Overall Survival
Description: Overall survival (OS) which was defined as the time from the date of randomisation to the date of death. Participants for whom there is no evidence of death at the time of the analysis will be censored at the date that they were last known to be alive.
Time Frame: From first drug administration until 28 days after last drug administration + Follow-Up period for collecting information on death, up to 2465 days.
Population: Randomised set which included all patients randomised to receive treatment, whether treated or not.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib | Gefitinib
Number analyzed (Participants) | 160 | 159
Months | 27.86 [25.13 to 32.85] | 24.54 [20.57 to 28.88]
Statistical Analysis 1: Comparison: Afatinib vs Gefitinib; Exploratory trial, no formal hypotheses were tested; Test type: Superiority or Other; p = 0.2343, Log Rank — p-value was not adjusted for multiple comparisons; Stratified by EGFR mutation group and presence of brain metastases at baseline; Hazard Ratio (HR) = 0.862, 95% CI 2-sided [0.674 to 1.101] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Objective Response Rate
Description: Objective response rate (ORR) which was defined as the number of participants with best overall response of complete response (CR) or partial response (PR) as assessed by central independent review according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1. divided by the total number of participants who received treatment. Per RECIST version 1.1. for target lesions and assessed by Computed Tomography (CT)-scan or Magnetic Resonance Imaging (MRI): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions from baseline. For the final analysis (analysis cut-off date 12 April 2019) objective response was determined by investigator assessment.
Time Frame: From first drug administration until 28 days after last drug administration + Follow-Up period for collecting information on disease progression, further anti-cancer treatment and death, up to 2465 days.
Population: Randomised set which included all patients randomised to receive treatment, whether treated or not.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib | Gefitinib
Number analyzed (Participants) | 160 | 159
Percentage of participants | 79.4 [72.3 to 85.4] | 74.8 [67.4 to 81.4]
Statistical Analysis 1: Comparison: Afatinib vs Gefitinib; Exploratory trial, no formal hypotheses were tested; Test type: Superiority or Other; p = 0.3235, Regression, Logistic — p-value was not adjusted for multiple comparisons; Stratified for EGFR mutation group and presence of brain metastases at baseline; Odds Ratio (OR) = 1.307, 95% CI 2-sided [0.768 to 2.223] — Ratio calculated as Afatinib divided by Gefitinib

5. Secondary Outcome: Time to Objective Response
Description: Number of participants with objective response (best overall response of complete response or partial response) to study treatment over time, cumulative number of participants is displayed. Time to objective response was defined as the time from randomisation to the first recorded objective response. For the final analysis (analysis cut-off date 12 April 2019) objective response was determined by investigator assessment.
Time Frame: as for outcome 4
Population: All participants in the randomised set with objective response.
Measure: Number; unit: Participants
Arm/Group | Afatinib | Gefitinib
Number analyzed (Participants) | 127 | 119
Participants
  Week 4 | 81 | 74
  Week 8 | 112 | 107
  Week 16 | 119 | 117
  Week 24 | 122 | 118
  Week 32 | 125 | 118
  Week 40 | 126 | 118
  Week 48 | 127 | 119

6. Secondary Outcome: Duration of Objective Response
Description: Duration of objective response defined as the time of first objective response (best overall response of complete response or partial response) to the time of progression or death, whichever occurred first (or date of censoring for progression free survival). For the final analysis (analysis cut-off date 12 April 2019) objective response was determined by investigator assessment.
Time Frame: as for outcome 4
Population: Participants in the randomised set with objective response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib | Gefitinib
Number analyzed (Participants) | 127 | 119
Months | 11.86 [10.12 to 15.54] | 11.07 [9.69 to 12.91]

7. Secondary Outcome: Disease Control
Description: Percentage of participants with disease control which was defined as the number of participants with best overall response of complete response (CR) or partial response (PR) or stable disease (SD) as assessed by central independent review according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1. divided by the total number of participants who received treatment. Per RECIST version 1.1. for target lesions and assessed by Computed Tomography (CT)-scan or Magnetic Resonance Imaging (MRI): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions from baseline; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Responses of SD were only considered if they occur ≥42 days from date of randomisation. For the final analysis (analysis cut-off date 12 April 2019) disease control was determined by investigator assessment.
Time Frame: as for outcome 1
Population: Randomised set which included all patients randomised to receive treatment, whether treated or not.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib | Gefitinib
Number analyzed (Participants) | 160 | 159
Percentage of participants | 94.4 [89.6 to 97.4] | 93.7 [88.7 to 96.9]
Statistical Analysis 1: Comparison: Afatinib vs Gefitinib; Exploratory trial, no formal hypotheses were tested; Test type: Superiority or Other; p = 0.7856, Regression, Logistic — p-value was not adjusted for multiple comparisons; Stratified for EGFR mutation group and presence of brain metastases at baseline; Odds Ratio (OR) = 1.138, 95% CI 2-sided [0.447 to 2.896] — Ratio calculated as Afatinib divided by Gefitinib

8. Secondary Outcome: Duration of Disease Control
Description: Duration of disease control defined as the time from randomisation to the time of progression or death, whichever occurred first (or date of censoring for progression free survival). For the final analysis (analysis cut-off date 12 April 2019) the status and date of disease progression were determined by investigator assessment.
Time Frame: as for outcome 1
Population: All participants in the randomised set with disease control, that is, with best overall response of complete response or partial response or stable disease.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib | Gefitinib
Number analyzed (Participants) | 151 | 149
Months | 12.88 [11.14 to 14.88] | 11.73 [10.58 to 14.55]

9. Secondary Outcome: Tumour Shrinkage (Main Overall Survival Analysis Cut-off Date, 08 April 2016)
Description: Tumour shrinkage assessed by minimum sum of post-baseline target lesion diameters recorded after randomisation. A positive value shows a decrease in tumour size.
Time Frame: From first drug administration until last drug administration, up to 1482 days
Population: Participants in the randomised set with tumour assessments.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimetre (mm)
Arm/Group | Afatinib | Gefitinib
Number analyzed (Participants) | 149 | 151
millimetre (mm) | 34.79 [32.18 to 37.40] | 38.25 [35.65 to 40.84]
Statistical Analysis 1: Comparison: Afatinib vs Gefitinib; Exploratory trial, no formal hypotheses were tested; Test type: Superiority or Other; p = 0.0657, ANCOVA — p-value was not adjusted for multiple comparisons; Adjusted for baseline sum of diameters, EGFR mutation group and presence of brain metastases at baseline; Mean Difference (Final Values) = -3.45, 95% CI 2-sided [-7.13 to 0.23], Standard Error of Mean 1.87 — Difference calculated as Afatinib minus Gefitinib

10. Secondary Outcome: Health-related Quality of Life (Primary Analysis Cut-off Date, 21 August 2015)
Description: Health-related quality of life (HRQoL) measured using European Quality of life - 5 Dimensions (EQ-5D) score for United Kingdom (UK) and Belgium and European European Quality Visual Analogue Scale (EQ-VAS).
  EQ-5D utility scores range from 0 (worst health) to 1 (full health).
  EQ-VAS scores range from 0 (worst imaginable health state) to 100 (best imaginable health state).
  Results display the mean score up to 56 weeks.
Time Frame: Every 8 weeks, up to 56 weeks
Population: All randomised subjects with health-related quality of life data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Afatinib | Gefitinib
Number analyzed (Participants) | 160 | 158
Units on a scale
  EQ-5D UK utility score | 0.77 [0.75 to 0.80] | 0.80 [0.77 to 0.82]
  EQ-5D Belgium utility score | 0.74 [0.72 to 0.77] | 0.77 [0.75 to 0.80]
  EQ-VAS utility score | 74.5 [72.3 to 76.6] | 76.0 [73.9 to 78.1]
Statistical Analysis 1: Comparison: Afatinib vs Gefitinib; EQ-5D UK utility score. Exploratory trial, no formal hypotheses were tested; Test type: Superiority or Other; p = 0.1422, Mixed Models Analysis — p-value was not adjusted for multiple comparisons; Adjusted for EGFR mutation group and presence of brain metastases at baseline; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.06 to 0.01], Standard Error of Mean 0.017 — Difference calculated as Afatinib minus Gefitinib
Statistical Analysis 2: Comparison: Afatinib vs Gefitinib; EQ-5D Belgium utility score. Exploratory trial, no formal hypotheses were tested; Test type: Superiority or Other; p = 0.0540, Mixed Models Analysis — p-value was not adjusted for multiple comparisons; Adjusted for EGFR mutation group and presence of brain metastases at baseline; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.06 to 0.00], Standard Error of Mean 0.016 — Difference calculated as Afatinib divided by Gefitinib
Statistical Analysis 3: Comparison: Afatinib vs Gefitinib; EQ-VAS utility score. Exploratory trial, no formal hypotheses were tested; Test type: Superiority or Other; p = 0.2032, Mixed Models Analysis — p-value was not adjusted for multiple comparisons; Adjusted for EGFR mutation group and presence of brain metastases at baseline; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-3.9 to 0.8], Standard Error of Mean 1.21 — Difference calculated as Afatinib divided by Gefitinib

ADVERSE EVENTS:
Time Frame: From first drug administration until 28 days after last drug administration, up to 2405 days. For All-Cause Mortality: From first drug administration until 28 days after last drug administration + Follow-Up period for collecting information on death, up to 2465 days.
Description: Treated set included all patients who were dispensed with and documented to have taken at least one dose of study medication. This set of patients was used for the evaluation of safety.
Arm/Group | Afatinib | Gefitinib
All-Cause Mortality (participants affected / at risk) | 126/160 | 132/159
Serious Adverse Events (participants affected / at risk) | 75/160 | 64/159
Other Adverse Events (participants affected / at risk) | 157/160 | 159/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (N=160) | Gefitinib (N=159)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 3
Cushing's syndrome (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 11 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3
Asthenia (General disorders) | 4 | 2
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 3
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Encephalitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 7 | 5
Sepsis (Infections and infestations) | 1 | 4
Skin bacterial infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Urosepsis (Infections and infestations) | 1 | 0
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 5
Dystonia (Nervous system disorders) | 1 | 0
Embolic cerebral infarction (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 3
Hydrocephalus (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1
Paraneoplastic encephalomyelitis (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 2
Confusional state (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Pneumonectomy (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Macular degeneration (Eye disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral disorder (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Large intestine infection (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (N=160) | Gefitinib (N=159)
Anaemia (Blood and lymphatic system disorders) | 14 | 5
Dry eye (Eye disorders) | 15 | 13
Abdominal pain (Gastrointestinal disorders) | 14 | 11
Abdominal pain upper (Gastrointestinal disorders) | 17 | 17
Constipation (Gastrointestinal disorders) | 29 | 24
Diarrhoea (Gastrointestinal disorders) | 143 | 102
Dry mouth (Gastrointestinal disorders) | 11 | 14
Dyspepsia (Gastrointestinal disorders) | 16 | 14
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 13
Mouth ulceration (Gastrointestinal disorders) | 20 | 7
Nausea (Gastrointestinal disorders) | 43 | 45
Stomatitis (Gastrointestinal disorders) | 63 | 18
Vomiting (Gastrointestinal disorders) | 31 | 19
Asthenia (General disorders) | 21 | 22
Chest pain (General disorders) | 20 | 19
Fatigue (General disorders) | 34 | 30
Influenza like illness (General disorders) | 3 | 8
Mucosal inflammation (General disorders) | 32 | 19
Oedema peripheral (General disorders) | 11 | 10
Pyrexia (General disorders) | 22 | 10
Conjunctivitis (Infections and infestations) | 14 | 10
Folliculitis (Infections and infestations) | 10 | 4
Nasopharyngitis (Infections and infestations) | 11 | 11
Paronychia (Infections and infestations) | 89 | 28
Upper respiratory tract infection (Infections and infestations) | 16 | 20
Urinary tract infection (Infections and infestations) | 18 | 9
Alanine aminotransferase increased (Investigations) | 19 | 44
Aspartate aminotransferase increased (Investigations) | 15 | 38
Weight decreased (Investigations) | 18 | 9
Decreased appetite (Metabolism and nutrition disorders) | 45 | 39
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 32
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 12
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 9 | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 | 17
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 10
Dizziness (Nervous system disorders) | 12 | 18
Headache (Nervous system disorders) | 14 | 22
Insomnia (Psychiatric disorders) | 13 | 9
Dysuria (Renal and urinary disorders) | 7 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 48 | 47
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 | 26
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 30 | 14
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 12 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 11 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 11
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 24 | 12
Acne (Skin and subcutaneous tissue disorders) | 5 | 17
Alopecia (Skin and subcutaneous tissue disorders) | 19 | 27
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 34 | 34
Dry skin (Skin and subcutaneous tissue disorders) | 52 | 63
Erythema (Skin and subcutaneous tissue disorders) | 10 | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 10 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 40 | 40
Rash (Skin and subcutaneous tissue disorders) | 100 | 87
Skin fissures (Skin and subcutaneous tissue disorders) | 23 | 6
Anxiety (Psychiatric disorders) | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.